CLINICAL TRIAL: NCT05133700
Title: Use and Opinions' Concerning Medicines Related Errors, Monitoring and Audit Tools Used to Assess Medicines Optimisation Within Care Homes in England
Brief Title: Use and Opinions of Care Home Medicines Audit Tools
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Malcolm Irons, Principal Investigator, University of Central Lancashire
Other Study IDs: HEALTH 0228CA; 280907 (Other: NHS Health Research Authority); 21/IEC08/0015 (Other: Social Care Research Ethics Committee)
Record Dates: First submitted 2021-10-15; First posted 2021-11-24 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Medication Systems; Quality Improvement
Keywords: Residential Facilities; Qualitative
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative interviews and focus group: Qualitative semi-structured individual interviews and focus groups to be held with people living in care homes (with and without nursing), health and social care staff supporting these people, commissioners and regulators.
  Interventions: Other: Interview or focus group discussion
- Qualitative medicines monitoring tools: Submission of current medicines monitoring tools by care homes and services supporting care homes including community pharmacies.
  Interventions: Other: Review of submitted medicines audit tools

INTERVENTIONS:
Other: Interview or focus group discussion — There is no intervention. This is a qualitative piece of work only
  Groups: Qualitative interviews and focus group
Other: Review of submitted medicines audit tools — There is no intervention. This is a qualitative piece of work only
  Groups: Qualitative medicines monitoring tools

SUMMARY:
To describe the barriers and facilitators experienced by residents, health and social care staff, commissioners and regulators when managing medicines within care homes.

DETAILED DESCRIPTION:
The prescribing of medicines is the most frequent health intervention in England. The administration or omission of medicines is not without risk and incidents involving medicines occur. The frequency of prescribing medicines increases with age and frailty. People living in care homes (with and without nursing) are generally older and more frail than similar groups in the community. Therefore, care homes and their staff need to be proficient and safe when administering medicines.

However, an under investigated area of prescribed medicines is the views of people living in care homes, health and social care staff, commissioners and regulator about managing medicines in care homes.

During the study a series of semi-structured interviews and focus groups will be undertaken. These focus groups will be held with people living in care homes (with and without nursing). Further interviews and focus groups will be held with health and social care staff, commissioners and regulators.

Care homes will be invited to provide copies of their current medicines monitoring tool. In addition, services supporting care homes including community pharmacies will also be invited to provide copies of their current medicines monitoring tools.

Analysis of conversations and monitoring tools made available to the study team will be undertaken and compared to published literature including grey literature.

ELIGIBILITY:
Inclusion Criteria:

1. Care homes

   * within pre-agreed areas,
   * registered with the regulator (CQC) for the regulated activities of Residential Care (with or without nursing) that have consented to participate.
   * Theses care homes will also be registered for one or more of the following specialisms:
   * dementia,
   * mental health conditions,
   * physical disabilities,
   * sensory impairments,
   * caring for adults under 65 years
   * caring for adults over 65 years.
2. Residents who have capacity and an adequate understanding of written and verbal English to consent and participate of participating care homes.
3. Care home staff, including registered managers who have an adequate understanding of written and verbal English to consent and participate of participating care homes.
4. Visiting health and social care staff who support care homes in the study locality.
5. Commissioner and regulatory staff with oversight of care homes in the study locality.
6. Medicines monitoring tools used by participating

   * care homes,
   * community pharmacies supporting the participating care homes
   * commissioners and regulators with oversight of care homes in the study locality.

Exclusion Criteria:

1. Care homes registered with the regulator (CQC)

   * outside of the pre-agreed areas.
2. Care homes registered with the regulator (CQC)

   * within the pre-agreed areas for the regulated activities of Residential Care (with or without nursing) that are also registered for the specialism of supporting younger people.
3. Residents of participating care homes judged by staff to lack capacity, an adequate understanding of written and verbal English to consent and participate, too unwell or might find it distressing.
4. Staff in participating care homes who lack an adequate understanding of written and verbal English to consent and participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Three geographical areas of England in different NHS regions
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators: qualitative semi-structured individual interviews | 0 to 9 months
  Transcribed interviews will be coded and then emerging themes from the data identified and developed. A constant comparison method of analysis will be used. The presence or lack of consensus and reinforcement on certain topics will also be observed.
Barriers and facilitators: qualitative semi-structured focus groups | 0 to 9 months
  Transcribed focus groups will be coded and then emerging themes from the data identified and developed. A constant comparison method of analysis will be used. The presence or lack of consensus and reinforcement on certain topics will also be observed.
Similarities and differences: current medicines monitoring tools | 9 to 12 months
  Current medicines monitoring tools will be coded and then emerging themes from the data identified and developed. A constant comparison method of analysis will be used. The presence or lack of consensus and reinforcement on certain topics will also be observed.
Qualitative comparative analysis | 9 to 12 months
  Themes and topics that emerged from the interviews, focus groups and current medicines monitoring tools will be compared and contrasted with each other and the evidence identified from a separate scoping review.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm W Irons, Principal Investigator — University of Central Lancashire
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No